CLINICAL TRIAL: NCT00494936
Title: HIV/HCV: Neuropsychiatric and Neurophysiological Features
Brief Title: Effects of HIV and Hepatitis C Virus on the Brain
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 03-0908; K23MH071181 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV; HCV; Treatment Naive; Treatment Experienced; HIV and HCV Coinfection
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HIV/HCV: HIV and HCV coinfected
- HIV infected: HIV monoinfected
- HIV/HCV nonviremnic: HIV and HCV coinfected with HCV RNA less than 600 copies
- HCV infected: HCV monoinfected with HCV viremia

SUMMARY:
This study will determine the effects that HIV and hepatitis C virus have on thinking abilities and whether the viruses affect brain chemistry.

DETAILED DESCRIPTION:
Hepatitis C is a liver disease that is caused by the hepatitis C virus (HCV). It can be successfully treated with 6 to 12 months of medication in both HIV infected and HIV uninfected people. Among HIV infected people, HCV infection is a common co-morbidity, and is more serious when it occurs in this population than others because it leads to liver damage more quickly. HIV is known to cause neurological deficits, and studies suggest that HCV may do so, as well. Knowledge about how to treat these deficits, however, is limited. More information about the nature of the neurological problems and their causes is needed to develop effective treatments. This study will determine the effects that HIV and HCV have on thinking abilities, such as memory, attention, and problem-solving, and whether the viruses affect brain chemistry.

Participants in this 4-year, observational study will undergo a series of tests and interviews. Participants may choose to complete all procedures over 2 days or three appointments. Procedures will include a 20-minute medical interview, a 4-hour neuropsychological evaluation, a 5-minute functional ability questionnaire, blood and urine collection (approximately 15 minutes), and a 1-hour magnetic resonance imaging (MRI) test of the head. The neuropsychological evaluation will test participants' memory, concentration, reasoning, and speed of thinking. All procedures will be completed over approximately 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* CD4 count is greater than 200
* Hepatitis C infected or uninfected
* Speaks English

Exclusion Criteria:

* Currently receiving interferon treatment for hepatitis C
* History of neurological illness
* Any psychotic spectrum disorder (e.g., schizophrenia or manic depression/bipolar disorder)
* History of learning disability
* History of head injury that entailed a loss of consciousness for more than 30 minutes
* Any metal in body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV / HCV Coinfected, HIV moninfected, & HCV monoinfected
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ryan, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Ryan EL, Morgello S, Isaacs K, Naseer M, Gerits P; Manhattan HIV Brain Bank. Neuropsychiatric impact of hepatitis C on advanced HIV. Neurology. 2004 Mar 23;62(6):957-62. doi: 10.1212/01.wnl.0000115177.74976.6c. PMID 15037699